CLINICAL TRIAL: NCT03116919
Title: Potatoes, Hypertension RIsk and Endothelial Function Study
Acronym: PHRIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lea Borgi, Associate Physician, Renal Division, Department of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000405
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Endothelial Dysfunction
Keywords: nutrition; Potatoes; endothelial function; feeding trial

STUDY DESIGN:
Intervention Model Description: Crossover feeding trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato arm (Other): One group will be fed an extra serving of boiled, baked or mashed potatoes daily for 1 week
  Interventions: Other: Potato
- Non-starchy vegetable (Other): Then crossover to an extra serving of a non-starchy vegetable
  Interventions: Other: Non-starchy vegetable

INTERVENTIONS:
Other: Potato — Participants will be given an extra serving of potato a day
  Arms: Potato arm
Other: Non-starchy vegetable — Participants will be given an extra serving of a non-starchy vegetable
  Arms: Non-starchy vegetable

SUMMARY:
White potatoes have recently been allowed back in the cash value voucher of the government food stamp program after it was stated that there were no known adverse health effects of potatoes. However, the association of potatoes with heart health, especially elevated blood pressure is not known. This study will examine the effects of potatoes on blood pressure in different populations of adults and children, and assess, in a feeding trial, the effects of an additional serving of potatoes per day on the possible mechanisms that link potatoes to high blood pressure. The investigators will also analyze the intake of potatoes in participants of the government food stamp program.

DETAILED DESCRIPTION:
Potatoes are one of the most consumed vegetables in the US and the world. In recent years, several changes have been made to government sponsored food programs with respect to potatoes, such as lifting the restriction on the number of servings of starchy vegetables (including potatoes) established by the Healthy Hunger-Free Act, and re-allowing white potatoes in the cash-value voucher for fruits and vegetables of the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC), after the Institute of Medicine asserted that there was insufficient evidence that white potatoes had adverse health effects. However, the investigators recently reported an increased incidence of hypertension with increasing potato consumption in three large prospective US cohort studies after adjusting for sodium intake and other potential confounders. The investigators also analyzed the association of short-term potato intake from a 24-hr dietary recall with endothelial-dependent vasodilation measured by brachial artery ultrasonography in the Modifiable Effectors of Renin System Activation Treatment Evaluation (MODERATE) trial. Participants who consumed one or more than one serving of boiled, baked or mashed potatoes during the previous day had a 1.7% lower endothelial-dependent vasodilation when compared with participants with no potato intake (p-value= 0.01) after adjusting for other factors. This is a relevant difference in endothelial function - by comparison, every 10 year increase in age was associated with a 1.2% lower endothelial function. Therefore, the investigators plan to analyze the effect of one serving of boiled, baked or mashed potato per day on endothelial function in a crossover feeding trial of healthy adult men and women.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* without known cardiovascular risk factor

Exclusion Criteria:

* History of hypertension, diabetes or cardiovascular disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function assessed by endothelium-dependent vasodilation using brachial artery ultrasonography | 1 week
  Change in endothelial function after eating potato or non-starchy vegetable

CONTACTS AND LOCATIONS:
Overall Officials: Lea Borgi, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided